CLINICAL TRIAL: NCT04992689
Title: Increasing Insulin Resistance as a Predictor of Impending Bacteremia: A Retrospective Study
Brief Title: Increasing Insulin Resistance as a Predictor of Impending Bacteremia
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr., Meir Medical Center
Other Study IDs: 0132-21-MMC
Record Dates: First submitted 2021-07-25; First posted 2021-08-05 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Acquired ICU Bacteremia
Keywords: acquired bacteremia, insulin resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Insulin resistance is defined as a decrease in the ability of insulin to lower blood glucose levels. Various pathological conditions can cause an increase in insulin resistance, such as sepsis, administration of certain medications, various stressful situations, surgery or significant injuries, etc. Sepsis can cause extreme stress, which causes significant changes in metabolism, disruption of blood glucose regulation and increased insulin resistance. In sepsis there is an extreme activation of inflammatory mediators and of counter-regulatory hormones, such as cortisol, glucagon and catecholamines, which increase hepatic gluconeogenesis on the one hand, and increase the peripheral resistance to insulin on the other hand.

Disorder in the regulation of blood glucose level causes increased mortality and morbidity among intensive care unit patients with sepsis, as well as an increase in the duration of hospitalization and its financial expenses.

There are a number of parameters used in the intensive care unit to diagnose the development of sepsis within the unit, such as an increase or decrease in body temperature, an increase in CRP level, white blood cell count, pro-calcitonin level, etc It is possible that an increase in insulin resistance can also be used as a predictor of sepsis. It should be noted that almost all patients hospitalized in the intensive care unit are treated with a continuous infusion of insulin to balance their blood glucose level, including patients who are not diagnosed with diabetes prior to their hospitalization in the unit. This is in light of the increase in insulin resistance for the reasons listed above among patients in critical condition, and also due to the need to maintain blood glucose values in the range of 140-180 mg/dl, since high blood glucose values among patients hospitalized in the intensive care unit are associated with increased morbidity and mortality.

We would therefore like to investigate whether an increase in insulin resistance, as expressed in an increase in the patient's insulin intake, can predict the development of sepsis secondary to bacteremia in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:Patients aged 18-100, diabetic and non-diabetic, admitted to the General Intensive Care Unit from January 2013 to January 2021 (inclusive) for any reason, required during their hospitalization a continuous infusion of insulin, and developed during their hospitalization acquired bacteremia after more than 48 hours from ICU admission.

-

Exclusion Criteria:Patients who did not receive a continuous insulin infusion, patients with bacteremia of non-pathogenic bacteria (contamination), patients who developed bacteremia less than 48 hours after ICU admission, patients who received drugs that might influence insulin resistance (steroids, glucagon) or patients with other reasons that might explain an increase in insulin resistance other than infection.

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acquired ICU bacteremia
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Increased insulin resistance as a predictor of impending ICU acquired bacteremia | 6 months post ICU admission
  To establish a possible connection between increasing insulin resistance, as measured by changes in insulin infusion rate (units per hour) in order to maintain blood glucose level between 140-180 mg%, and development of acquired ICU bacteremia (at least 48 hours post ICU admission)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Dichtwald, Dr, Principal Investigator — Meir Medical Center
Locations (1):
- Meir medical center Kfar Saba, Kfar Saba, Israel